CLINICAL TRIAL: NCT01097161
Title: The Speech Prosody of People With Stuttering and Developmental Apraxia: the Efficacy of an Intervention Program
Brief Title: Stuttering and Apraxia of Speech: the Efficacy of an Intervention Program
Acronym: SAS:EIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Bernadette von Atzingen Santos Cardoso, Laboratório de Fonética -UFMG
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHA 0097/06
Record Dates: First submitted 2010-03-31; First posted 2010-04-01 (Estimated); Last update posted 2010-04-02 (Estimated); Status verified 2007-04

CONDITIONS: Stuttering; Developmental Apraxia of Speech
Keywords: Stuttering; Apraxia of speech; Motor control; Prosody; Pitch range; Speech rate; fluency disorders
MeSH Terms: conditions — Stuttering; Apraxias | interventions — Speech Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Speech treatment on prosodic basis (Experimental): Patients receive 20 therapy sessions over a course of 3 months, with one double session per week.
  Interventions: Behavioral: speech therapy with the assistance of an acoustical analysis program

INTERVENTIONS:
Behavioral: speech therapy with the assistance of an acoustical analysis program — Two weekly speech sessions realized on individual basis for three months period

SUMMARY:
Subjects' utterances were submitted to acoustic analysis before and after the intervention program applied on prosodic basis.

DETAILED DESCRIPTION:
The study has the aim of developing knowledge, methodology and technique in the prosody area, for its application on the speech therapy, with the assistance of a feedback system - with WinpitchPro (Philippe Martin). A database was constituted on the basis of a patterned corpus (EUROM1) by its translation, recording and editing on .wav format. Throughout model-sentences, an experimental intervention program initiates with the participation of 2 adults with stuttering problem and 2 with apraxia of speech. The efficacy of the therapeutic procedure is tested on the basis of the acoustical and the statistical analyses which have compared the first and the second speech samples taken before and after the twenty (20) therapy sessions held in a prosody approach only.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of stuttering
* Clinical diagnosis of apraxia of speech
* 18 years of age or older
* Portuguese native language
* Agreement by the participant to enroll on 20 therapy sessions scheduled in a 3 month period

Exclusion Criteria:

* History of major medical illness unrelated to primary diagnosis of developmental stuttering and developmental apraxia of speech
* Significant abnormalities on general physical and neurological examination unrelated to primary diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2007-04; Primary Completion 2007-10 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- R. Grão Pará, 85/404, Belo Horizonte, Minas Gerais, Brazil

REFERENCES:
- See also: Laboratório de Fonética da FALE - UFMG — http://www.letras.ufmg.br/labfon
- See also: Conselho nacional de Saúde — http://portal2.saude.gov.br/sisnep/pesquisador
- See also: Fundação de Amparo à pesquisa do Estado de Minas Gerais — http://www.fapemig.br